CLINICAL TRIAL: NCT00040768
Title: A Phase II Study Of PS-341 In Metastatic Non-Small Cell Lung Cancer
Brief Title: Bortezomib in Treating Patients With Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02470; UPCC 06501; CDR0000069405 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who received prior bortezomib and achieved at least a partial response of at least 6 months duration may also receive therapy as above.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Phase II trial to study the effectiveness of bortezomib in treating patients who have stage IIIB, stage IV, or recurrent non-small cell lung cancer. Bortezomib may interfere with the growth of tumor cells by blocking certain enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, time to progression, and survival of patients with advanced non-small cell lung cancer treated with bortezomib.

II. Determine the toxicity of this drug in these patients. III. Correlate toxicity and activity of this drug with markers of proteasome inhibition in blood and peripheral mononuclear cells in these patients.

OUTLINE:

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who received prior bortezomib and achieved at least a partial response of at least 6 months duration may also receive therapy as above.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Mixed tumors allowed unless small cell elements are present
* Stage IIIB or IV or recurrent disease
* At least 1 measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastases
* Performance status - ECOG 0-1
* More than 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver involvement present)
* Creatinine ≤ 2 mg/dL
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy > grade 1
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No more than 1 prior chemotherapy regimen

  * Two prior chemotherapy regimens allowed provided 1 of the 2 regimens was gefitinib monotherapy as second-line therapy
* At least 4 weeks since prior chemotherapy (6 weeks for carmustine, mitomycin, or nitrosoureas) and recovered
* At least 4 weeks since prior radiotherapy (except localized radiotherapy for symptom relief) and recovered
* Prior bortezomib allowed provided patient achieved at least a partial response (of at least 6 months duration), received no other therapy since the last dose of bortezomib, and has no residual toxicity greater than grade 1
* No other concurrent investigational or commercial agents or therapies for malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-04; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate to PS-341 therapy | Up to 4 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 4 months
  Kaplan-Meier estimates of survival (overall, progression free) and 95% confidence intervals will be calculated.
Overall survival | Up to 4 hours
  Kaplan-Meier estimates of survival (overall, progression free) and 95% confidence intervals will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: James Stevenson, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States